CLINICAL TRIAL: NCT03755804
Title: Pediatric Classical Hodgkin Lymphoma Consortium Study: cHOD17
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: Teva Pharmaceuticals USA (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: cHOD17; NCI-2018-02924 (Registry Identifier: NCI Clinical Trial Registration Program)
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Hodgkin Lymphoma
Keywords: Hodgkin Lymphoma; Pediatric Cancer; Frontline Therapy; Response Adapted Therapy; Risk Adapted Therapy
MeSH Terms: conditions — Hodgkin Disease; Neoplasms | interventions — Bendamustine Hydrochloride; Etoposide; Doxorubicin; Bleomycin; Vincristine; Vinblastine; Prednisone; Prednisolone; Filgrastim; Brentuximab Vedotin; Cyclophosphamide; Dacarbazine; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low-Risk (Experimental): Participants receive 2 cycles of BEABOVP: bendamustine, etoposide, Adriamycin® (doxorubicin), bleomycin, Oncovin® (vincristine), vinblastine and prednisone. Filgrastim may be given as clinically indicated. Dexrazoxane may be given at the discretion of the treating investigator. Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an AR after 2 cycles of therapy. Quality of Life measurements may be done.
  Interventions: Drug: bendamustine; Drug: Etoposide; Drug: Doxorubicin; Drug: Bleomycin; Drug: Vincristine; Drug: Vinblastine; Drug: Prednisone; Drug: Filgrastim; Other: Quality of Life Measurements; Radiation: Radiotherapy
- Intermediate-Risk (Experimental): Participants receive 3 cycles of BEABOVP: bendamustine, etoposide, Adriamycin® (doxorubicin), bleomycin, Oncovin® (vincristine), vinblastine and prednisone. For patients with an AR after 2 cycles of therapy, steroids will be omitted from their subsequent cycles of therapy. Filgrastim may be given as clinically indicated. Dexrazoxane may be given at the discretion of the treating investigator. Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an AR after 2 cycles of therapy. Quality of Life measurements may be done.
  Interventions: Drug: bendamustine; Drug: Etoposide; Drug: Doxorubicin; Drug: Bleomycin; Drug: Vincristine; Drug: Vinblastine; Drug: Prednisone; Drug: Filgrastim; Other: Quality of Life Measurements; Radiation: Radiotherapy
- High-Risk (Experimental): Participants receive 2 cycles of AEPA: Adcedris® (brentuximab vedotin), etoposide, prednisone and Adriamycin® (doxorubicin) and 4 cycles of CAPDac: cyclophosphamide, Adcetris® (brentuximab vedotin), prednisone and Dacarbazine® (DTIC). For patients with an AR after 2 cycles of therapy, steroids will be omitted from their subsequent cycles of therapy. Filgrastim may be given as clinically indicated. Dexrazoxane may be given at the discretion of the treating investigator. Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an AR after 2 cycles of therapy. Quality of Life measurements may be done.
  Interventions: Drug: Etoposide; Drug: Doxorubicin; Drug: Prednisone; Drug: Filgrastim; Drug: Brentuximab Vedotin; Drug: Cyclophosphamide; Drug: DTIC; Other: Quality of Life Measurements; Radiation: Radiotherapy

INTERVENTIONS:
Drug: bendamustine — Given intravenously (IV)
  Other Names: TREANDA (R)
  Arms: Intermediate-Risk; Low-Risk
Drug: Etoposide — Given intravenously (IV)
  Other Names: VP-16; Vepeside
Drug: Doxorubicin — Given intravenously (IV)
  Other Names: Adriamycin (R)
Drug: Bleomycin — Given intravenously (IV)
  Other Names: Blenoxane (R)
  Arms: Intermediate-Risk; Low-Risk
Drug: Vincristine — Given intravenously (IV)
  Other Names: Oncovin (R)
  Arms: Intermediate-Risk; Low-Risk
Drug: Vinblastine — Given intravenously (IV)
  Other Names: Velban (R)
  Arms: Intermediate-Risk; Low-Risk
Drug: Prednisone — Given orally (PO)
  Other Names: Prednisolone
Drug: Filgrastim — Given subcutaneously (SQ) or IV
  Other Names: Neupogen (R)
Drug: Brentuximab Vedotin — Given intravenously (IV)
  Other Names: Adcetris
  Arms: High-Risk
Drug: Cyclophosphamide — Given intravenously (IV)
  Other Names: Cytoxan (R)
  Arms: High-Risk
Drug: DTIC — Given intravenously (IV)
  Other Names: DACARBAZINE (R); Dimethyl Triazeno Imidazole Carboximide
  Arms: High-Risk
Other: Quality of Life Measurements — Quality of Life measurements may be done in low-risk cycles 1 and 2 BEABOVP, intermediate-risk cycles 1, 2 and 3 BEABOVP and high-risk cycles 1 and 2 AEPA and cycles 1, 2, 3, and 4 CAPDac. QOL may be done at year 1, 2 and 5 for all risk groups.
  Other Names: Quality of Life Measurements (QOL)
Radiation: Radiotherapy — Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an AR after 2 cycles of therapy for all risk groups. Radiotherapy will be administered after completion of all chemotherapy upon hematologic count recovery.
  Other Names: radiation therapy; irradiation

SUMMARY:
This is a phase II study using risk and response-adapted therapy for low, intermediate and high risk classical Hodgkin lymphoma. Chemotherapy regimens will be based on risk group assignment. Low-risk and intermediate- risk patients will be treated with bendamustine, etoposide, Adriamycin® (doxorubicin), bleomycin, Oncovin® (vincristine), vinblastine, and prednisone (BEABOVP) chemotherapy. High-risk patients will receive Adcetris® (brentuximab vedotin), etoposide, prednisone and Adriamycin® (doxorubicin) (AEPA) and cyclophosphamide, Adcetris® (brentuximab vedotin), prednisone and Dacarbazine® (DTIC) (CAPDac) chemotherapy. Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an adequate response (AR) after 2 cycles of therapy for all risk groups.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

* To evaluate the efficacy (adequate response) after 2 cycles of BEABOVP (bendamustine substitution for mechlorethamine in the original Stanford V chemotherapy backbone) in low-risk and intermediate-risk patients with classical Hodgkin lymphoma (cHL).
* To estimate the event-free survival in high-risk patients with classical Hodgkin lymphoma (cHL).

SECONDARY OBJECTIVES

* To describe the acute hematologic and infectious toxicities of BEABOVP (bendamustine substitution for mechlorethamine in the original Stanford V chemotherapy backbone) in patients with low-risk and intermediate- risk cHL as they relate to transfusion requirements, hematopoietic growth factor support, episodes of febrile neutropenia and hospitalizations, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
* To describe the acute hematologic, neuropathic, and infectious toxicities of AEPA/CAPDac in patients with high-risk cHL as they relate to transfusion requirements, hematopoietic growth factor support, episodes of grade 3 and 4 sensory or motor neuropathy, episodes of febrile neutropenia and hospitalizations, according to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
* To evaluate patterns of failure in irradiated and non-irradiated patients.
* To estimate the EFS functions of LR and IR patients, and compare with those in previously published studies.
* To estimate the response rate in HR patients and compare with historical and literature rates.
* To compare response rates in LR and IR patients with historical and literature rates.
* To compare the EFS function of HR patients with that in previously published studies.

EXPLORATORY OBJECTIVES

* To evaluate the plasma pharmacokinetics of bendamustine along with predictors of its variability when used as part of BEABOVP regimen for pediatric cHL patients
* To explore the patterns and dynamics of T-cell clonality in classical Hodgkin lymphoma
* To explore the association between TARC, total metabolic tumor volume, stage, risk group and treatment response.
* To establish next generation sequencing of ctDNA as a reliable method of non-invasively profiling tumor-associated mutations in pediatric patients with HL.
* To determine if kinetics of ctDNA in patients with pediatric HL during treatment are predictive of outcome.
* To obtain baseline testing by St. Jude Lifetime Study (SJLIFE) to allow for enhanced survivorship follow-up:

  * Neurologic testing
  * Neurocognitive testing
  * Quantitative brain imaging
  * Polysomnography
  * Cardiovascular testing (valvular testing, arterial elasticity, carotid-femoral pulse wave velocity, orthostatic hypotension, heart rate variability
  * Neuropathy screening
  * Changes in body mass index composition during therapy

Low-risk and Intermediate-risk: Low-risk patients will receive 2 cycles of BEABOVP and Intermediate-risk patients will receive 3 cycles of BEABOVP.

BEABOVP regimen: Patients will receive bendamustine day 1, etoposide day 15, Adriamycin® (doxorubicin) days 1 and 15, bleomycin days 8 and 22, Oncovin® (vincristine) days 8 and 22, vinblastine days 1 and 15, and prednisone two or three times per day every other day of each cycle for a total of 14 days of steroids.

High-risk patients will receive 2 cycles of AEPA and 4 cycles of CAPDac.

AEPA regimen: Patients will receive Adcedris® (brentuximab vedotin) days 1, 8 and 15, etoposide days 1 to 5, prednisone two or three times daily days 1 to 15 and Adriamycin® (doxorubicin) days 1 and 15.

CAPDac regimen: Patients will receive cyclophosphamide days 1 and 8, Adcetris® (brentuximab vedotin) days 1 and 8, prednisone two or three times daily days 1 to 15 and Dacarbazine® (DTIC) days 1 to 3.

Residual node radiotherapy will be given at the end of all chemotherapy only to involved nodes that do not have an AR after 2 cycles of therapy for all risk groups.

Steroids will be omitted after 2 cycles for any IR or HR patient with an AR after 2 cycles of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, previously untreated CD30+ classical HL. (Participants are still eligible if they received limited emergent RT or steroid therapy - maximum of 7 days if within the last month or as approved by PI).
* Age ≤ 21 years at the time of diagnosis (i.e., participants are eligible until their 22nd birthday) for low-risk and intermediate-risk
* Age ≤ 25 years at the time of diagnosis (i.e., participants are eligible until their 26th birthday) for high-risk
* All Ann Arbor stages.

  * Low-Risk: IA, IIA (excluding patients with "E" lesions or mediastinal bulk)
  * Intermediate-Risk: IA or IIA with "E" lesions or bulky mediastinal adenopathy (mediastinal mass to thoracic cavity ratio 33% or greater by chest radiograph) and IB, IIIA.
  * High-Risk: IIB, IIIB, IV
* Adequate renal function based on GFR ≥ 70 ml/min/1.73m2 OR serum creatinine adjusted for age and gender as follows: Age 1 to < 2 years: maximum serum creatinine 0.6 mg/dL for males and 0.6 mg/dL for females, Age 2 to < 6 years: maximum serum creatinine 0.8 mg/dL for males and 0.8 mg/dL for females, Age 6 to < 10 years: maximum serum creatinine 1 mg/dL for males and 1 mg/dL for females, Age 10 to < 13 years: maximum serum creatinine 1.2 mg/dL for males and 1.2 mg/dL for females, Age 13 to < 16 years: maximum serum creatinine 1.5 mg/dL for males and 1.4 mg/dL for females, Age ≥16 years: maximum serum creatinine 1.7 mg/dL for males and 1.4 mg/dL for females
* Adequate hepatic function (total bilirubin ≤ 1.5 x ULN for age, and AST/ALT ≤ 2.5 x ULN for age).
* Adequate hematologic criteria at baseline, unless secondary to Hodgkin disease diagnosis

  * Absolute neutrophil count (ANC) ≥1000/µL
  * Platelets ≥ 75,000/µL
* Adequate cardiac function defined as shortening fraction of ≥ 27% by echocardiogram or MUGA, unless decreased function is due to large mediastinal mass or effusion related to HL.
* Adequate pulmonary function defined as no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 92% on room air unless secondary to a large mediastinal mass or effusion related to HL.
* Female participant who is post-menarchal must have a negative urine or serum pregnancy test.
* Female or male participant of reproductive potential must agree to use an effective contraceptive method throughout duration of study treatment.

Exclusion Criteria:

* CD30 negative HL.
* Has received prior therapy for Hodgkin lymphoma
* Inadequate organ function
* High-risk participants with a history of ≥ grade 2 peripheral neuropathy or any active neurologic disease that would impede the ability to assess neurologic toxicities.
* Inability or unwillingness of research participant or legal guardian / representative to give written informed consent.

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 232 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Response rate of adequate response | after the first 2 cycles of chemotherapy (at approximately 2 months after enrollment
  The 70 evaluable low-risk patients enrolled will be evaluated for this objective.
Response rate of adequate response | after the first 2 cycles of chemotherapy (at approximately 2 months after enrollment
  The 65 evaluable intermediate-risk patients enrolled will be evaluated for this objective
Event-free survival | From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment
  Time to event defined as relapse, progression or death. The 115 evaluable high-risk patients participants enrolled will be evaluated for this objective.

SECONDARY OUTCOMES:
Number of adverse events in low-risk and intermediate-risk patients | From enrollment to end of therapy (approximately 8 months
  According to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Number of adverse events in high-risk patients | From enrollment to end of therapy (approximately 8 months
  According to the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0
Local failure rate | From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment
  Local failure rate in irradiated and non-irradiated patients
Event-free survival | From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment
  Time to event defined as relapse, progression or death. The EFS for the low-risk patients and intermediate-risk patients are compared to those in HOD08 and HOD05, respectively.
Response rate | after the first 2 cycles of chemotherapy (at approximately 2 months after enrollment
  Response rate of adequate response after 2 cycles of AEPA in the high-risk patients with FDG-PET compared to that after 2 cycles of AEPA in HLHR13.
Response rate | after the first 2 cycles of chemotherapy (at approximately 2 months after enrollment
  Response rate of adequate response after 2 cycles of BEABOVP in the low-risk and high-risk patients with FDG-PET compared to those after 2 cycles of STANFORD V chemotherapy in HOD08 and HOD05, respectively.
Event-free survival | From start of therapy to 2 years after completion of therapy (up to 3 years after study enrollment
  Time to event defined as relapse, progression or death. The EFS for the high-risk patients is compared to those in HLHR13.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Ehrhardt, MD, MS, Principal Investigator — St. Jude Children's Research Hospital
Locations (8):
- United States (8):
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - St. Jude Midwest Affiliate - Peoria, Peoria, Illinois
  - St. Jude Affiliate Baton Rouge Clinic (Our Lady of the Lakes Regional Medical Center), Baton Rouge, Louisiana
  - Maine Children's Cancer Program, Scarborough, Maine
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - St. Jude Affiliate Clinic at Novant Health Hemby Children's Hospital, Charlotte, North Carolina
  - St. Jude Children's Research Hospital, Memphis, Tennessee

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: ClinicalTrials Open at St. Jude — http://www.stjude.org/protocols